CLINICAL TRIAL: NCT03613363
Title: Engineering Evaluation of the Helix Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Respironics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HRC-17067-HCPED-CC
Record Dates: First submitted 2018-07-09; First posted 2018-08-03 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Disease; Pulmonary Disease; Pediatric ALL
MeSH Terms: conditions — Respiration Disorders; Lung Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: This trial is an engineering study is to verify the overall performance and controls of the Helix Ventilator as compared to the participant's current therapy device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Helix Ventilator (Experimental): The Helix ventilator is a non-FDA cleared ventilator device. The Helix ventilator has similar modalities to the Trilogy ventilator, which has FDA clearance. The Helix device has improved algorithms, controls, and features to enhance the therapy delivery. Additionally, Helix has an updated hardware platform which has been adequately tested to ensure that the device specifications are met. No pre-clinical or developmental clinical work was required because of Trilogy being the established predicate.
  Interventions: Device: Helix Ventilator

INTERVENTIONS:
Device: Helix Ventilator — The Helix ventilator is a non-FDA cleared ventilator device. The Helix ventilator has similar modalities to the Trilogy ventilator, which has FDA clearance. The Helix device has improved algorithms, controls, and features to enhance the therapy delivery. Additionally, Helix has an updated hardware platform which has been adequately tested to ensure that the device specifications are met. No pre-clinical or developmental clinical work was required because of Trilogy being the established predicate.

SUMMARY:
This study will be used to evaluate and observe the overall performance and controls of the Helix ventilator. Pressure and flow data between participants' current devices and the Helix ventilator will be assessed in either invasive or non-invasive ventilation. To evaluate ventilator performance, pressure and waveform data will be assessed as well. Also, patient and caregiver feedback will be captured. The target population is infants to adults weighing more than 5kg. Participants will be recruited by Boston Children's Health Physician's Group. Up to thirty participants will be enrolled in the study.

DETAILED DESCRIPTION:
Following the completion of the informed consent, participants enrolled in this study will be asked to use their existing ventilator for up to 1 hour to collect pressure and flow data for comparison purposes against the Helix ventilator.

Participants will then be set up on the Helix Ventilatory System using the same mode of therapy as their current ventilator. Participants may receive mechanical ventilation using any patient circuit currently being designed for the Helix Ventilator (Passive, Active with Positive Airway Pressure (PAP), Active with Flow, or dual limb). Patients currently using non-invasive ventilation may be asked to use a mouth piece in lieu of a mask interface. While using the study device, therapy setting may be altered by the physician or his/her surrogate while maintaining the ventilator needs of the patient. For e.g.,a patient currently prescribed an synchronized intermittent mechanical ventilation (SIMV) mode may temporarily be switched to a pressure control mode to assess patient synchrony and ventilator performance.

Once the participant is set-up, he/she will be asked to use the ventilator for up to 4 hours. During this time, Philips Respironics engineers will be collecting data through several mechanisms: 1) Helix SanDisc (SD) Card, 2) Non-invasive Cardiac Output (NICO) Monitoring System, and / or 3) External data collection device (ex. laptop). The study staff may ask the participant's opinions on the comfort of the therapy delivery. There will be no invasive monitoring as part of this study.

The engineering evaluations will take place at the Boston Children's Health Physician offices. The study investigators, respiratory therapist, and/or other qualified clinical staff, will be supervising and present for all study visits. Philips Respironics engineers will be present for observational purposes only. All study staff working on this trial will be trained to the protocol and device prior to beginning work.

Participants may be asked to participate in this data collection study up to six (6) times.

Study data collected for this study will be collected on paper or electronic source records. These records will include information regarding inclusion/exclusion, performed study procedures and questions regarding device use. Only those staff that have been delegated by the Principal Investigator will be able to enter or make changes to the data in the Case Report Forms.

ELIGIBILITY:
Inclusion Criteria:

Participants who are currently using mechanical ventilation (> 1 month at time of study participation) as part of medical care and have demonstrated a clinically acceptable response to this therapy and meet the following inclusion criteria:

1. Weight > 5Kg;
2. Any medical condition requiring mechanical ventilation through nasal/facial mask, mouthpiece or tracheostomy
3. Any medical condition requiring mechanical ventilation for > 1 month

Exclusion Criteria:

1. Participants intubated with an endotracheal tube
2. Clinically unstable, i.e.,

   1. Acute Respiratory Failure
   2. Participants with refractory hypotension (defined as systolic blood pressure less than 90 mm Hg despite inotropic agents)
   3. Uncontrolled cardiac ischemia or arrhythmias d. Any participant determined as inappropriate for the study by the Principal Investigator
3. Patients suffering from metastatic or terminal cancer
4. Currently employed by a manufacturer of respiratory products or family member employed by a manufacturer of respiratory products
5. Patient of surrogate is unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- New York Medical College, Hawthorne, New York, United States

IPD SHARING:
Plan to Share IPD: No
All data will stay within Philips.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Helix Ventilator
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Evaluable Population: This population of non-invasive patients completed the engineering evaluation and utilized settings that allowed proper comparison between Trilogy and their current ventilator.
- Non-Evaluable Population: This population included N=2 invasive-ventilator patients, as well as N=1 who did not complete the engineering evaluation, and N=4 who were only included for the purposes of testing the updated leak algorithm.
- Total: Total of all reporting groups
Arm/Group | Evaluable Population | Non-Evaluable Population | Total
Number analyzed (Participants) | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.3 (10.2) | 16.3 (8.5) | 13.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 11 | 4 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 7 | 20

OUTCOME MEASURES:

1. Primary Outcome: Proximal Pressure From Trilogy Evo Ventilator and Current Device
Description: Proximal pressure from the participant's Trilogy Evo ventilator and current device
Time Frame: 1 day
Population: This population of non-invasive patients completed the engineering evaluation and utilized settings that allowed proper comparison between Trilogy and their current ventilator. It excludes N=2 invasive-ventilator patients, as well as N=1 who did not complete the engineering evaluation, and N=4 who were only included for the purposes of testing the updated leak algorithm.
Measure: Mean (Standard Deviation); unit: cm H2O
Groups:
- Evaluable Population: Trilogy Evo: Proximal Pressure (cm H2O) while on Trilogy Evo therapy
- Evaluable Population: Current Device: Proximal Pressure (cm H2O) while using current device
Arm/Group | Evaluable Population: Trilogy Evo | Evaluable Population: Current Device
Number analyzed (Participants) | 13 | 13
cm H2O | 8.3 (1.6) | 8.2 (3.0)

2. Primary Outcome: Proximal Flow From Trilogy Evo and Patient's Current Device
Description: Proximal flow from Trilogy Evo and patient's current device
Time Frame: 1 day
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters / minute
Groups:
- Evaluable Population: Trilogy Evo: Proximal Flow (L/min) while on Trilogy Evo therapy
- Evaluable Population: Current Device: Proximal Flow (L/min) while using current device
Arm/Group | Evaluable Population: Trilogy Evo | Evaluable Population: Current Device
Number analyzed (Participants) | 13 | 13
Liters / minute | 4.2 (4.5) | 4.9 (5.7)

3. Secondary Outcome: Subjective Ease-of-Operation Rating Regarding Trilogy Device
Description: Subjective Ease-of-Operation rating (1-Very Easy to 5-Very Hard) regarding Trilogy device
Time Frame: 1 day
Population: This population of non-invasive patients completed the engineering evaluation and utilized settings that allowed proper comparison between Trilogy and their current ventilator. It excludes N=2 invasive-ventilator patients, as well as N=1 who did not complete the engineering evaluation, and N=4 who were only included for the purposes of testing the updated leak algorithm. Data not available from N=1 participant.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Ease of Operation: Trilogy Evo: Trilogy Evo therapy
Arm/Group | Ease of Operation: Trilogy Evo
Number analyzed (Participants) | 12
scores on a scale | 1.9 (0.8)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Helix Ventilator
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/63/NCT03613363/Prot_SAP_000.pdf